CLINICAL TRIAL: NCT01948258
Title: Clearblue Advanced Fertility Monitor Consumer One Cycle at Home Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SPD Development Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 0481
Record Dates: First submitted 2013-09-18; First posted 2013-09-23 (Estimated); Results first posted 2018-11-02 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2018-01

CONDITIONS: Pregnancy
Keywords: Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Clearblue Advanced Fertility Monitor (Other): Use of Clearblue Fertility Monitor
  Interventions: Device: Clearblue Advanced Fertility Monitor

INTERVENTIONS:
Device: Clearblue Advanced Fertility Monitor — Clearblue Advanced Fertility Monitor used for one menstrual cycle in a home setting

SUMMARY:
This study will assess the use of the new Clearblue Advanced Fertility Monitor for one menstrual cycle in a home setting by female volunteers seeking to get pregnant.

DETAILED DESCRIPTION:
The Clearblue Fertility Monitor is a personal monitor designed to be used with disposable test sticks for the semi-quantitative measurement of estrone-3-glucuronide (E3G) and luteinising hormone (LH) in women's urine. This personal information allows women to identify their fertile window and appropriately time intercourse in order to maximise their chances of conception. A new version of this monitor (Clearblue Advanced Fertility Monitor) has been developed with additional functionality including the option to test for pregnancy.

This study will assess the volunteer ease of use of the new Clearblue Advanced Fertility Monitor and the understanding and interpretation of the results by the user. This is a single centre clinical study which will be conducted by volunteers at their residence and co-ordinated by the clinical department at SPD Development Company Ltd.

A minimum of 100 female volunteers representing the target consumer will be required to use the new Clearblue Advanced Fertility Monitor at home as per the instructions for use. This will involve them setting up the monitor, using the monitor for one full cycle and then setting up the monitor for their next cycle unless they test for pregnancy and get a pregnant result.

At the end of one full cycle, all volunteers will complete a study questionnaire which includes sections on comprehension of the instructions for use, ease of use and interpretation of test results.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Aged 18 - 45 years
* Willing to provide written informed consent to participate in the study and comply to the investigational procedures
* Naive to similar marketed products including current Clearblue fertility monitor and Persona
* Two natural cycles immediately prior to entering the study, each lasting between 21 and 42 days
* Seeking to become pregnant

Exclusion Criteria:

* Unwilling to provide written informed consent to participate in the study or comply with study procedures
* Employees of SPD, Proctor & Gamble or Alere
* Have a condition that is known to be contra-indicated in pregnancy
* Usually have menstrual cycles which are shorter than 21 days or longer than 42 days
* Using or have used in their last 2 cycles, hormonal contraceptives including oral, emergency oral, implants, patches, transdermal injections, vaginal ring and progesterone intrauterine systems (IUS)
* Using or have used in the last 2 cycles, infertility medications or hormone replacement therapy containing hCG or LH
* Taking clomiphene citrate or other ovulation induction drugs
* Are using any treatment which may affect the menstrual cycle
* Have recently been pregnant, miscarried or breastfeeding
* Have been diagnosed with polycystic ovarian syndrome (PCOS)
* Are peri- or post-menopausal e.g. experiencing symptoms such as irregular menstrual periods, hot flushes, night sweats, sleep disturbances and mood swings
* Are taking antibiotics containing tetracyclines
* Have impaired liver or kidney function
* Have previously participated in a SPD 'trying to conceive' study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 395 (Actual)
Dates: Start 2013-03-01; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Johnson, PhD, Study Director — SPD Swiss Precision Diagnostics GmbH
Locations (1):
- SPD Development Company Ltd, Bedford, Bedfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Overall results will be shared after study completion

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted by volunteers remotely and managed by the clinical department at SPD. For the study, 395 females aged between 18-45 years were recruited via internet advertising and from women who had participated in previous SPD studies. The first volunteer was recruited on 1st March 2013, the last was recruited on 1st August 2013.
Pre-assignment Details: Volunteers were instructed to test for pregnancy prior to starting the study. If pregnant before the start of their cycle they were withdrawn and classified as a pre-study pregnancy. Volunteers were also withdrawn if identified as health care professionals.
Groups:
- Fertility Monitor: Use of Clearblue Advanced Fertility Monitor
Period: Overall Study
Arm/Group | Fertility Monitor
Started | 395
Completed | 233
Not Completed | 162
Not completed — Pregnancy | 41
Not completed — Did not complete by cut-off date | 35
Not completed — Lost to Follow-up | 27
Not completed — Withdrawal by SPD | 8
Not completed — Withdrawal by Subject | 6
Not completed — Health Care Professional | 43
Not completed — Removed from statistical analysis | 2

BASELINE CHARACTERISTICS:
Population: All volunteers recruited
Groups:
- Fertility Monitor: Use of Clearblue Fertility Monitor
Arm/Group | Fertility Monitor
Number analyzed (Participants) | 233
Age, Customized [Count of Participants; unit: Participants] — Age of Participants who used the new Clearblue Advanced Fertility Monitor
  Participants
    Age of Participants: 18-25 | 38
    Age of Participants: 26-30 | 68
    Age of Participants: 31-35 | 64
    Age of Participants: 36-40 | 56
    Age of Participants: 41-45 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 233
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Asian : Bangladeshi | 0
  Race/Ethnicity: Asian : Chinese | 3
  Race/Ethnicity: Asian : Indian | 3
  Race/Ethnicity: Asian : Pakistani | 6
  Race/Ethnicity: Asian : South Asian | 0
  Race/Ethnicity: Asian : Other Asian | 2
  Race/Ethnicity: Black: African | 3
  Race/Ethnicity: Black: Caribbean | 1
  Race/Ethnicity: Black: Other Black | 1
  Race/Ethnicity: Native Hawaiian or other Pacific Islander | 0
  Race/Ethnicity: American Indian or Alaska Native | 0
  Race/Ethnicity: White: American | 3
  Race/Ethnicity: White: Australian/New Zealander | 0
  Race/Ethnicity: White: Eastern European | 0
  Race/Ethnicity: White: Mediterranean/Middle Eastern | 0
  Race/Ethnicity: White: Western European | 210
  Race/Ethnicity: White: Other White | 1
  Race/Ethnicity: Mixed | 0
Highest qualification [Count of Participants; unit: Participants]
  Post-graduate qualifications | 25
  Degree or equivalent (college degree) | 77
  Other higher education below degree level (associa | 20
  A levels, vocational level 3 and equivalents (age | 55
  GCSE (Grade A*-C), vocational level 2 and equivale | 41
  Qualifications at level 1 and below | 2
  Other qualifications | 8
  No qualifications | 5
Occupation [Count of Participants; unit: Participants]
  Managerial | 23
  Professional | 59
  Associate Professional / Technical | 27
  Administrative / Secretarial | 24
  Skilled Trade | 4
  Personal Services | 8
  Sales / Customer Services | 29
  Manufacturing / Driver | 0
  Support Personnel | 11
  Student | 4
  Homemaker | 32
  Other | 12

OUTCOME MEASURES:

1. Primary Outcome: The Ability of the Volunteer to Use the New Clearblue Advanced Fertility Monitoring a Home Setting
Description: Acceptance criteria is that ≥80% of volunteers will score 3 or less on the Likert scale in a home setting by demonstrating ease of use and comprehension of the instructions for use.
Time Frame: one month use
Population: Volunteers whose data contributes to the full analysis set.
Measure: Number; unit: percentage of participants
Arm/Group | Fertility Monitor
Number analyzed (Participants) | 233
percentage of participants | 89.7

2. Secondary Outcome: Correct Identification of Monitor Status
Description: To demonstrate correct user identification of fertility status and test days and to determine the performance of the monitor in consumer hands.
Time Frame: one month
Population: Volunteers who completed the study, who had daily diary entries and monitor download data for days on which a test was conducted
Measure: Number; unit: percentage of participants
Arm/Group | Fertility Monitor
Number analyzed (Participants) | 228
percentage of participants | 91.2

3. Other Pre Specified Outcome: Pregnancy Test Result
Description: Pregnancy test results will also be compared with both the performance of a currently marketed pregnancy test when used by a trained technician and quantitative hCG concentration.
Time Frame: one month
Population: Volunteers who completed the study, comparison of Clearblue Fertility Monitor pregnancy test results and a marketed pregnancy test. Results for all tests conducted.
Measure: Number (95% Confidence Interval); unit: percentage of tests in agreement
Arm/Group | Fertility Monitor
Number analyzed (Participants) | 329
percentage of tests in agreement
  Monitor test result in agreement with predicate | 99.3 [97.6 to 99.9]
  Monitor test result in agreement with hCG levels | 100 [98.8 to 100]

ADVERSE EVENTS:
Time Frame: Duration of study, one cycle per volunteer.
Arm/Group | Fertility Monitor
All-Cause Mortality (participants affected / at risk) | 0/393
Serious Adverse Events (participants affected / at risk) | 0/393
Other Adverse Events (participants affected / at risk) | 0/393

LIMITATIONS AND CAVEATS:
There was some incomplete data with women not using the monitor on all the days that ideally would have been tested. We believe the missing data did not affect the objectives of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes